CLINICAL TRIAL: NCT03722095
Title: The Effects of Preconditioning Theta Burst Stimulation With Transcranial Direct Current Stimulation on Stress Regulation in Healthy Controls: a Double-blind Sham-controlled Study
Brief Title: Research on the Effects of Combined Neurostimulation Protocols on Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: EC/2018/0866
Record Dates: First submitted 2018-10-02; First posted 2018-10-26 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Stress Reaction; Stress Related Disorder; Major Depressive Disorder
Keywords: Non-invasive Brain Stimulation; intermittent Theta Burst Stimulation (iTBS); Transcranial Direct Current Stimulation (tDCS); Dorsolateral Prefrontal Cortex; Stress reactivity; Stress-related Disorders; Major Depressive Disorder
MeSH Terms: conditions — Fractures, Stress; Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS + active iTBS (Active Comparator): Participants will receive 20 minutes of active tDCS, during the last 7 minutes active iTBS will be applied.
  Interventions: Device: active tDCS; Device: iTBS
- sham tDCS + active iTBS (Sham Comparator): Participants will receive 20 minutes of sham tDCS, during the last 7 minutes active iTBS will be applied.
  Interventions: Device: sham tDCS; Device: iTBS

INTERVENTIONS:
Device: active tDCS — A current of 2 milliampère (mA) through electrodes of 5x5cm.
  Other Names: active/anodal transcranial direct current stimulation
  Arms: active tDCS + active iTBS
Device: sham tDCS — Similar set-up as in the active tDCS, but stimulation is too short to cause any effects.
  Other Names: sham transcranial direct current stimulation
  Arms: sham tDCS + active iTBS
Device: iTBS — 54 cycles with 10 bursts of 3 pulses, train duration of 2 seconds and intertrain intervals of 6 seconds, results in 1620 pulses at 110% resting motor threshold.
  Other Names: intermittent theta burst stimulation

SUMMARY:
The study examines the effects of the combined use of two different non-invasive brain stimulation (NIBS) techniques targeting the DLPFC on stress reactivity and recovery.

DETAILED DESCRIPTION:
Transcranial Direct Current Stimulation (tDCS) will be combined with intermittent Theta Burst Stimulation (iTBS) in order to maximize the effects coming from each of the techniques on their own. A group of 74 healthy participants wil be submitted to two different stimulation protocols (sham tDCS + active iTBS and active tDCS + active iTBS) with one-week in between and results on stress reactivity will be examined. In order to improve therapeutic protocols, this study with healthy participants is a crucial first step in order to further conduct clinical studies with psychiatric samples.

ELIGIBILITY:
Inclusion Criteria:

- Aged between 18-45 years old

Exclusion Criteria:

* The presence of psychiatric disorders
* Usage of psychotropic medication
* Any or cardiovascular neurological condition
* Personal or family history of epilepsy or other neurological disorders
* Unstable medical condition, as well as chronic pain conditions, (such as fibromyalgia) or increased blood pressure
* Eye disease(s)
* Current substance abuse
* Inner ear prosthesis
* Any implanted electronic device susceptible for magnetic field radiation (e.g. pacemaker)
* Any implanted metal device in the head region
* Metal objects or magnetic objects in the brain or around the head (only removable earrings & piercing are allowed)
* Recent neurosurgical interventions
* Pregnancy
* Skin problems in the head region
* Recent fractures or wounds on the hand

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate variability (HRV) | Through study completion, an average of two weeks
  Variability in time between two heartbeats

SECONDARY OUTCOMES:
Changes in heart rate (HR) | Through study completion, an average of two weeks
  Beats per minute
Changes in blood pressure (BP) | Through study completion, an average of two weeks
  Both systolic and diastolic blood pressure (SBP/DBP)
Changes in electrodermal activity (EDA) | Through study completion, an average of two weeks
  Peak amplitudes of Skin Conductive Responses (SCRs)
Changes in state-dependent mood | Through study completion, an average of two weeks
  Visual analogue scales (VAS): total scores will be reported (range 0 to 10) with higher scores indicating worse outcome
Changes in state-dependent ruminative thinking | Through study completion, an average of two weeks
  Brief State Rumination Inventory (BSRI): total scores will be reported (range 0 to 80) with higher scores indicating worse outcome
Changes in anxiety features - self-report | Through study completion, an average of two weeks
  State/Trait Anxiety Inventory (STAI): total scores will be reported (range 0 to 160) with higher scores indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Chris Baeken, MD, PhD, Principal Investigator — Ghent University, University Hospital Ghent; Marie-Anne Vanderhasselt, PhD, Principal Investigator — Ghent University, University Hospital Ghent; Stefaan Van Damme, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be made public on the open science framework website.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After study completion.
Access Criteria: Open acces
URL: https://osf.io